CLINICAL TRIAL: NCT00877630
Title: Minimal Invasiveness of Endoscopic Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Second Military Medical University (Other)
Responsible Party: Ming Qiu/Minimally Invasive Surgical Center, Changzheng Hospital affiliated to SMMU
Other Study IDs: SMMU-2-2009-2
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1:endoscopic group: patients underwent endoscopic thyroidectomy
- 2:conventional group: patients underwent open thyroidectomy

SUMMARY:
The investigators had performed more than 250 cases of breast approach endoscopic thyroidectomy (BAET). The goal of this study is to evaluate whether BAET could be a minimally invasive procedure under the expert's hands.

ELIGIBILITY:
Inclusion Criteria:

* thyroidectomy nodule diagnosed by ultrasound

Exclusion Criteria:

* thyroid carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients admitted in the ward who are diagnosed with thyroid nodule and will undergo thyroidectomy
Sampling Method: Non-Probability Sample
Dates: Start 2006-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Serum IL-6 and CRP levels before and after operation | 0, 2, 12, 24, 48 hours after surgery
Visual Analogue Scale (VAS) score | 2, 12, 24, 48 hours after surgery
Cosmetic outcomes after surgery | 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ming Qiu, MD., Ph D, Study Director — SMMU
Locations (1):
- Minimally Invasive Surgical Center of Changzhang Hospital, Shanghai, China